CLINICAL TRIAL: NCT02940171
Title: Impact of Timing of Surgery on Outcome of Severely Ill Burn Patients
Brief Title: Timing of Surgery And Outcome in Burn Patients ( EARLYBURN )
Acronym: EARLYBURN
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI 14029
Record Dates: First submitted 2016-10-17; First posted 2016-10-20 (Estimated); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Burns
Keywords: burns; critically ill; surgery outcome; mortality
MeSH Terms: conditions — Burns; Critical Illness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and urine bank 1 / day of inclusion (D0): 1 sample (3 x 5 ml of blood). 1 sample (10 ml sample of urine) 2 / The seventh day of inclusion (D7): 1 sample (3 x 5 ml of blood) 1 sample (10 ml sample of urine) 3 / The twenty eighth day of inclusion (D28): 1 sample (3 x 5 ml of blood) 1 sample (10 ml sample of urine) 4 / The sixtieth day of inclusion (J60) or the day of the release from hospital: 1 sample (3 x 5 ml of blood) 1 sample (10 ml sample of urine) The aliquots will be stored locally at -20 °C or 80°C Every 6 months, they will be transported to the "Centre de Ressources Biologiques" (CRB) of the Lariboisière Hospital. The samples will be preserved for 10 years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Early surgery: Early Excision of full thickness burn First excision surgery of full -thickness burn performed within 48 hours from burn injury
  Interventions: Procedure: Early Excision of full thickness burn
- Late surgery: Late Excision of full thickness burn First excision surgery of full -thickness burn performed after 48 hours from burn injury
  Interventions: Procedure: Late Excision of full thickness burn

INTERVENTIONS:
Procedure: Early Excision of full thickness burn — first excision surgery of full -thickness burn performed within 48 hours from burn injury
  Other Names: Early
  Groups: Early surgery
Procedure: Late Excision of full thickness burn — first excision surgery of full -thickness burn performed after 48 hours from burn injury
  Other Names: Late
  Groups: Late surgery

SUMMARY:
The prognostic of burn patients has improved over the last decades. Early excision of full thickness burns is thought to be one of the key factors which have led to prognostic improvement. Best timing for burn excision remain uncertain, however. In this multicenter observational study, we aim at exploring the impact of timing of surgery on outcome in severely ill burn patients using a propensity analysis.

DETAILED DESCRIPTION:
The first aim of the study is to explore the impact of timing of the first surgery on outcome of severely ill burn patients. Because a randomization would not be feasible in this setting, we will use a propensity analysis in matching patients receiving early surgery and those receiving late surgery. Secondary aims are to evaluate the impact of the timing of surgery on morbidity (organs failure, infections, sepsis) but also to assess the diagnostic and prognostic value of plasma and urine biomarkers in severely ill burn patients

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Admission to a burn unit within 72 hours from a burn injury
* Total burned surface area (TBSA)>20%(2nd degree or 3rd degree) for any type of burn
* Patient covered by the social security
* Non-opposition to participate to the study and to the constitution of the biological collection

Exclusion Criteria:

* Decline to participate
* Decision not to resuscitate order before surgery
* Pregnant or breastfeeding patiente
* Decision to limit therapies in the first 24 hours
* Patient not resident in France
* Patient deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with extensive skin burns, defined as greater than 20% of the total body surface
Sampling Method: Probability Sample
Enrollment: 470 (Actual)
Dates: Start 2016-12-25 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
mortality | 90 days

SECONDARY OUTCOMES:
Organ failure | 28 and 60 days
Recovery from acute kidney | Until 28 and 60 days from burn injury
Median Sequential Organ Failure Assessment score (SOFA score) during first 28 days | First 28 days
  Median Sequential Organ Failure Assessment score (SOFA score) during first 28
Nosocomial infections (numbers) during first 60 days | First 60 days
  Nosocomial infections (numbers) during first 60 days
Nosocomial sepsis during first 60 days | First 60 days
  Nosocomial sepsis during first 60 days
Length of stay in the ICU | One year
  Length of stay in the ICU
analog scale of quality of life | One year
  Functional sequel at one year, the patient will assesassess his overall quality of life since his accident Scale 1 to 10, with 1: poor, 10: good
One year mortality | One year
  One year mortality

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu Dr Legrand, MD, PhD, Principal Investigator — Saint-Louis Hospital, Paris, France; Mourad BENYAMINA, MD, PH, Principal Investigator — Saint-Louis Hospital, Paris, France
Locations (1):
- Departement of Anesthesiology, Critical Care and Burn Unit; Saint-Louis hospital, University Paris Diderot, Paris, France

IPD SHARING:
Plan to Share IPD: No